CLINICAL TRIAL: NCT05172960
Title: Safety and Effectiveness of Balloon-Expandable Bioprosthetic SAPIEN X4 Transcatheter Heart Valve
Brief Title: ALLIANCE: Safety and Effectiveness of the SAPIEN X4 Transcatheter Heart Valve
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-05
Record Dates: First submitted 2021-12-14; First posted 2021-12-29 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Aortic Stenosis, Severe
Keywords: Transcatheter aortic valve replacement (TAVR); Transcatheter aortic valve implantation (TAVI); SAPIEN X4
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TAVR - Main Cohort (Experimental): Subjects will undergo transcatheter aortic valve replacement (TAVR)
  Interventions: Device: SAPIEN X4 THV
- TAVR - Bicuspid Registry (Experimental): Subjects with bicuspid aortic valve morphology will undergo TAVR
  Interventions: Device: SAPIEN X4 THV

INTERVENTIONS:
Device: SAPIEN X4 THV — Implantation of the SAPIEN X4 valve

SUMMARY:
The objective of this study is to establish the safety and effectiveness of the Edwards SAPIEN X4 Transcatheter Heart Valve (THV) in subjects with symptomatic, severe, calcific aortic stenosis (AS).

DETAILED DESCRIPTION:
This is a prospective, single arm, multicenter study. Subjects with bicuspid aortic valve morphology will be enrolled in a separate registry.

ELIGIBILITY:
Inclusion Criteria:

1. Severe, calcific AS
2. Native aortic annulus size suitable for SAPIEN X4 THV
3. NYHA functional class ≥ II
4. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Anatomical characteristics that would preclude safe femoral placement of the introducer sheath or safe passage of the delivery system
2. Aortic valve is unicuspid, bicuspid or non-calcified
3. Pre-existing mechanical or bioprosthetic valve in any position
4. Severe aortic regurgitation (> 3+)
5. Severe mitral regurgitation (> 3+) or ≥ moderate mitral stenosis
6. Need for mitral, tricuspid or pulmonic valve intervention within the next 12 months
7. Left ventricular ejection fraction < 20%
8. Cardiac imaging evidence of intracardiac mass, thrombus or vegetation
9. Left ventricular outflow tract calcification that would increase the risk of annular rupture or significant PVL after THV implantation
10. Increased risk of coronary artery obstruction after THV implantation
11. Myocardial infarction within 30 days prior to the study procedure
12. Hypertrophic cardiomyopathy with subvalvular obstruction
13. Subjects with planned concomitant ablation for atrial fibrillation
14. Complex coronary artery disease (CAD) that cannot be optimally treated by percutaneous coronary intervention (PCI)
15. Any surgical or transcatheter procedure within 30 days prior to the study procedure (unless part of planned strategy for treatment of CAD). Implantation of a permanent pacemaker or implantable cardioverter defibrillator (ICD) is not considered an exclusion.
16. Any planned surgical or transcatheter intervention to be performed within 30 days following the study procedure (unless part of planned strategy for treatment of CAD)
17. Endocarditis within 180 days prior to the study procedure
18. Stroke, transient ischemic attack or neurological signs and symptoms attributed to carotid or vertebrobasilar disease within 90 days prior to the study procedure
19. Hemodynamic or respiratory instability requiring inotropic or mechanical support within 30 days prior to the study procedure
20. Renal insufficiency and/or renal replacement therapy
21. Leukopenia, anemia, thrombocytopenia
22. Inability to tolerate or condition precluding treatment with antithrombotic therapy
23. Hypercoagulable state or other condition that increases risk of thrombosis
24. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with premedication
25. Subject refuses blood products
26. BMI > 50 kg/m2
27. Estimated life expectancy < 24 months
28. Female who is pregnant or lactating
29. Active SARS-CoV-2 infection or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments
30. Participating in another investigational drug or device study that has not reached its primary endpoint
31. Subject considered to be part of a vulnerable population

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 915 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Non-hierarchical composite of death and stroke | 1 year
  The number of patients that died or had a stroke

SECONDARY OUTCOMES:
Favorable outcome per VARC-3: Composite of 1) alive, 2) Kansas City Cardiomyopathy Questionnaire (KCCQ) score ≥ 60, and 3) KCCQ score decrease ≤10 points from baseline | 1 year
  The number of patients that met all of these criteria. The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Paravalvular leak | 30 days
  Paravalvular leak will be categorized as None, Trace, Mild, Mild-Moderate, Moderate, Moderate-Severe, or Severe
New permanent pacemaker implantation | 30 days
  The number of patients with this event

CONTACTS AND LOCATIONS:
Overall Officials: Tamim M. Nazif, MD, Principal Investigator — Columbia University; Rahul P. Sharma, MBBS, Principal Investigator — Stanford University
Locations (65):
- United States (58):
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Kaiser Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UC Davis Medical Center Sacramento, Sacramento, California
  - Bay Area Structural Heart at Sutter Health, San Francisco, California
  - Kaiser San Francisco Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - UC Health Northern Colorado (Medical Center of the Rockies), Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Naples Community Hospital Healthcare System, North Naples, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Atlanta, Atlanta, Georgia
  - Rush University Medical Center Chicago, Chicago, Illinois
  - Alexian Brothers Hospital Network, Elk Grove Village, Illinois
  - NorthShore University HealthSystem Research Institute Evanston, Evanston, Illinois
  - Northwestern University Chicago, Evanston, Illinois
  - Silver Cross Hospital, New Lenox, Illinois
  - St. Vincent Medical Group, Inc./ St. Vincent Heart Center of Indiana, LLC, Carmel, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Washington University - Barnes-Jewish Hospital Saint Louis, St Louis, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Dartmouth-Hitchcock Medical Center, Hanover, Lebanon, New Hampshire
  - Atlantic Health System Morristown, Morristown, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - University at Buffalo - Kaleida Health, Buffalo, New York
  - Cornell Medical Center, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Montefiore Medical Center, New York, New York
  - Carolinas Health System, Charlotte, North Carolina
  - Novant Health and Heart Vascular Institute, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Cardiovascular Research Group Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Kaiser Portland, Clackamas, Oregon
  - Providence Heart & Vascular Institute Portland, Portland, Oregon
  - Pinnacle Health Harrisburg, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Methodist Le Bonheur Healthcare, Germantown, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Saint Thomas Health, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - University of Texas Memorial Hermann, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington Seattle, Seattle, Washington
- Australia (3):
  - St. Andrews War Memorial Hospital, Spring Hill, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Royal Melbourne Hospital, Parkville
- Canada (3):
  - St. Paul's Hospital System, Vancouver, British Columbia
  - Hamilton Health Services, Hamilton, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec- Universite Laval, Québec, Quebec
- Christchurch Hospital, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No